CLINICAL TRIAL: NCT05606302
Title: A Multi-center Clinical Study of Drug Antibody and Precision Transfusion in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2019-164
Record Dates: First submitted 2022-11-02; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-06

CONDITIONS: Drug-specific Antibodies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Piperacillin group: Blood samples for hemolytic anemia in patients treated with piperacillin were screened for the production of drug antibodies.
- Amoxicillin group: Blood samples for hemolytic anemia in patients treated with amoxicillin were screened for the production of drug antibodies.
- Cefazolin group: Blood samples for hemolytic anemia in patients treated with cefazolin were screened for the production of drug antibodies.
- Cefuroxime group: Blood samples for hemolytic anemia in patients treated with cefuroxime were screened for the production of drug antibodies.
- Ceftriaxone group: Blood samples for hemolytic anemia in patients treated with ceftriaxone were screened for the production of drug antibodies.
- Cefoxitin sodium group: Blood samples for hemolytic anemia in patients treated with cefoxitin sodium were screened for the production of drug antibodies.
- Vancomycin group: Blood samples for hemolytic anemia in patients treated with vancomycin were screened for the production of drug antibodies.

SUMMARY:
Blood samples for hemolytic anemia in patients treated with one or more of the antibiotics including piperacillin, amoxicillin, cefazolin, cefuroxime, ceftriaxone, cefoxitin sodium, and vancomycin were screened for the production of drug antibodies.

DETAILED DESCRIPTION:
The widespread use of antibiotics and anti-tumor drugs in clinical practice leads to poor efficacy or even toxic side effects and other adverse events, which are often related to the immune response caused by the cells adsorption or binding because of the long-term use of drugs to cause the generation of antibodies or drug decomposition.The immune hemolytic anemia caused by antibiotics is more common.In this study, the remaining blood samples of patients who developed hemolytic anemia using one or more antibiotics including piperacillin, amoxicillin, cefazolin, cefuroxime, ceftriaxone, cefoxitin sodium and vancomycin were preliminarily screened to determine which drugs caused hemolytic anemia.The types of diseases and antibiotics used in patients with drug-induced hemolytic anemia were also analyzed.The positive rate of drug antibody production was calculated and the difference of drug antibody production mechanism was analyzed.The blood samples of the positive patients and some negative patients were collected and preserved to prepare for the follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent;
* No limitation on age or sex;No limitation on nationality;Regional unlimited;
* Participates treated with one or more of the drugs including piperacillin, amoxicillin, cefazolin, cefuroxime, ceftriaxone, cefoxitin sodium, and vancomycin.

Exclusion Criteria:

* High fat blood sample;
* Sample of severe hemolysis;
* Jaundice sample;
* The sample is cloudy and may be contaminated with bacteria;
* The source of the sample is unknown and cannot be traced;
* Patients with a history of medication who were deemed inappropriate to participate in this study were evaluated by the researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with one or more of the antibiotics including piperacillin, amoxicillin, cefazolin, cefuroxime, ceftriaxone, cefoxitin sodium, and vancomycin.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To compare the positive rate of drug antibody between different drugs. | through study completion, an average of 3 years.
  The drug-induced hemolytic anemia test kit (microcolumn gel method) was used to determine whether drug antibodies were produced in the participates.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital of southern medical university, Guangzhou, Gaungdong, China